CLINICAL TRIAL: NCT03224715
Title: Actinic Cheilitis Pre-Treated With DNA Repair Enzyme Cream
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project was withdrawn and never began at Loyola University Medical Center.
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Rebecca Tung, Director of Dermatology, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 210079
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Actinic Cheilitis
MeSH Terms: conditions — Actinic cheilitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Actinic Cheilitis patients (Experimental)
  Interventions: Other: DNA Repair Enzyme Cream

INTERVENTIONS:
Other: DNA Repair Enzyme Cream — ver-the-counter cosmeceutical. We were going to be using it adjunctively before standard treatment of the actinic cheilitis was done

SUMMARY:
It is well known that ultraviolet (UV) light causes sunburn and DNA damage that can lead to skin cancer. Despite preventative measures of sunscreens and other topicals the incidence of skin cancers continues to increase every year. Chronic exposure can lead to development of both basal and squamous cell carcinoma that also is correlated to the risk of melanoma. When epidermal keratinocytes are exposed to UV radiation, they form cyclobutane pyrimidine dimmers (CPDs), 6-pyrimidine-4-pyrimidones (6-4-PPs), and oxygen radicals that alter the structure of nucleotides. When these lesions are not repaired, DNA replication is altered that leads to mutations in p53 and PTCH tumor suppressor gene and ultimately tumor development. It has been discovered that intracellular delivery of bacterial DNA incision repair enzyme T4 endonuclease V DNA repair enzymes can repair sun induced damaged DNA in patients with xeroderma pigmentosum4,. Yarosh et al also showed that T4 endonuclease V DNA repair enzymes are specific to reducing the amount of cyclobutane pyrimidine dimers and were found to lower the rate of new actinic keratoses compared to placebo lotion by 68% with no adverse effects observed. Additionally Yarosh et al also showed that T4N5 liposomes can repair keratinocyte DNA in skin cancer patients. This study will examine if pretreating actinic cheilitis with DNA repair enzyme cream before standard treatments can decrease the need for additional and possibly more aggressive therapies, decrease the surface area of affected areas, and possibly improve skin thickening and texture.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with clinically confirmed actinic cheilitis
* Fitzpatrick Type I, II, III, or IV skin.
* At least 20% of upper and/or lower lip affected by actinic cheilitis

Exclusion Criteria:

* Pregnant or nursing
* Allergies to any component of the study topical medication
* Prior treatment of actinic cheilitis within the past month, including cryotherapy, PDT, 5-FU, Picato, Retinoid, Diclofenac
* Prior ablative laser therapy to the lips, including fractional erbium and CO2 lasers.
* Prior use of lip fillers
* Presence of any skin disease that might interfere with the study treatments, including, but not limited to, rosacea, atopic dermatitis, lip lickers dermatitis, perioral dermatitis, perleche, active herpes infection.
* Presence of hypertrophic and hyperkeratotic lesions or cutaneous horns within the treatment area
* Any diagnosis of active, untreated skin cancer of the lip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of complete clearance vs partial response, determined clinically and by high-resolution macrophotography through blinded dermatologist evaluation | 12 weeks
  Percentage of patients with no clinically visible remaining lesions in treated area For partial responders: differentiate approximate surface area of affected lips, expressed as a percentage (0 to 100), compared with that prior to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola Dermatology, La Grange Park, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Berker D, McGregor JM, Hughes BR; British Association of Dermatologists Therapy Guidelines and Audit Subcommittee. Guidelines for the management of actinic keratoses. Br J Dermatol. 2007 Feb;156(2):222-30. doi: 10.1111/j.1365-2133.2006.07692.x. PMID 17223860
- [Background] Yarosh D, Klein J, O'Connor A, Hawk J, Rafal E, Wolf P. Effect of topically applied T4 endonuclease V in liposomes on skin cancer in xeroderma pigmentosum: a randomised study. Xeroderma Pigmentosum Study Group. Lancet. 2001 Mar 24;357(9260):926-9. doi: 10.1016/s0140-6736(00)04214-8. PMID 11289350
- [Background] Mouret S, Baudouin C, Charveron M, Favier A, Cadet J, Douki T. Cyclobutane pyrimidine dimers are predominant DNA lesions in whole human skin exposed to UVA radiation. Proc Natl Acad Sci U S A. 2006 Sep 12;103(37):13765-70. doi: 10.1073/pnas.0604213103. Epub 2006 Sep 5. PMID 16954188
- [Background] Cleaver JE. Defective repair replication of DNA in xeroderma pigmentosum. 1968. DNA Repair (Amst). 2004 Feb 3;3(2):183-87. PMID 15344228